CLINICAL TRIAL: NCT04391140
Title: Effectiveness of Prone Positioning Combined With High-flow Nasal Cannula for Patients With COVID-19 Induced ARDS
Brief Title: Prone Positioning and High-flow Nasal Cannula in COVID-19 Induced ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AG)198/2020
Record Dates: First submitted 2020-05-10; First posted 2020-05-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-05

CONDITIONS: COVID; ARDS; Acute Respiratory Distress Syndrome; Acute Respiratory Failure; Corona Virus Infection
Keywords: PRONE POSITION; High flow nasal cannula
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Combination of prone position and HFNC
  Interventions: Other: Prone position
- Control (No Intervention): Standard care: HFNC set for a SpO2 90-95% if unless indication for intubation is present.

INTERVENTIONS:
Other: Prone position — HFNC set to a SpO2 of 90-95% combined with prone position. At least 2 sessions of 30 minutes or more will be performed daily.
  Arms: Experimental

SUMMARY:
Prone position (PP) has been proved to be effective in severe ARDS patients. On the other hand, High flow nasal cannula (HFNC) may prevent intubation in hypoxemic Acute respiratory failure (ARF) patients.

Our hypothesis is that the combination of PP and HFNC in patients with COVID19 induced ARDS may decrease the need of mechanical ventilation.

Primary outcome: Therapeutic failure within 28 days of randomization (death or intubation). Secondary outcomes: to analyze PP feasibility and safety in HFNC patients and to analyze effectiveness in terms of oxygenation.

Methods: multicentric randomized study including patients with COVID19 induced ARDS supported with HFNC. Experimental group will received HFNC and PP whereas observation group will received standard care.

Optimization of non-invasive respiratory management of COVID19 induced ARDS patients may decrease the need of invasive mechanical ventilation and subsequently ICU and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 pneumonia according to the diagnostic criteria in effect at the time of inclusion or very strongly suspected.
* Patient treated by nasal high flow.
* Moderate or severe ARDS: bilateral radiological opacities not explained entirely by effusions, atelectasis or nodules; acute hypoxemia with worsening within the 7 previous days, not entirely explained by left ventricular failure; PaO2 / FiO2 ratio <300 mmHg (or SpO2 / FiO2 equivalent).
* Informed consent.
* Beneficiary or affiliated to a social security scheme.

Exclusion Criteria:

* Indication of immediate tracheal intubation
* Significant acute progressive circulatory insufficiency
* Impaired alertness, confusion, restlessness
* Body mass index> 40 kg / m2
* Chest trauma or other contraindication to prone position
* Pneumothorax
* Vulnerable person: safeguard of justice
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Therapeutic failure death or intubation | 28 days within randomization
  Therapeutic failure: death or intubation

SECONDARY OUTCOMES:
Feasibility and safety of prone position in HFNC patients | 28 days within randomization
  1. Comfort measurement using a visual-analog scale.
  2. Presence of complications related with prone position and the use of high-flow nasal cannula:
     1. Skin ulcers.
     2. Intravascular lines displacement
     3. HFNC related events (hot air feeling, nasal lesions)
Efficacy of prone position in HFNC patients | 28 days within randomization
  1. Evolution of the oxygenation (SpO2/FiO2) in prone position.
  2. Efficacy
     1. Length of HFNC therapy
     2. Length of ICU stay
     3. Length of mechanical ventilation (in those who require intubation)
     4. ICU and hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared to perform a meta-trial including other studies that assess the effectiveness of prone position in COVID-19 patients supported with nasal high flow.
  No patient identifying data will be transferred to the data repository. The data set will use pseudoanonymised data. The consent process for the study will highlight that this is a meta-trial and that both aggregated and individual data without personal identifying features will be used to formulate the results from the study. Local regulation for the management of patient data needs to be adhered to as part of agreement for involvement in the study.
  Data will be shared during the study at two points, Time 1 An interim analysis at 200 patients in which aggregated outcome data for the primary outcome and severe adverse effects will be analyzed
  Time 2 Final analysis outlining salient clinical feature of patients for each group, outcomes
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared when first 200 patients (counting the 5 studies participating in the meta-trial) will be included and at the end of inclusion

REFERENCES:
- [Derived] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Derived] Tavernier E, McNicholas B, Pavlov I, Roca O, Perez Y, Laffey J, Mirza S, Cosgrave D, Vines D, Frat JP, Ehrmann S, Li J. Awake prone positioning of hypoxaemic patients with COVID-19: protocol for a randomised controlled open-label superiority meta-trial. BMJ Open. 2020 Nov 11;10(11):e041520. doi: 10.1136/bmjopen-2020-041520. PMID 33177145